CLINICAL TRIAL: NCT02150408
Title: Evaluation of PET-CT Using Somatostatin Agonists Labeled With Gallium68 in Neuroendocrine Tumors
Acronym: DOTATATENET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-27
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Gastro-Entero-Pancreatic Tumors (GEPs)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- assesment by 68Ga-DOTATATE PET-CT (Experimental)
  Interventions: Other: PET-CT

INTERVENTIONS:
Other: PET-CT

SUMMARY:
Gastro-Entero-Pancreatic tumors (GEPs) are a subset of Neuroendocrine tumors (NETs) derived from the primitive gut and include digestive and bronchial NETs.

Historically, the gold standard in their functional exploration is the "conventional" somatostatin receptors scintigraphy (SRS) labeled with Indium-111 (Octreoscan®). This reference imaging is complementary to Tomography (CT) and liver MRI. However SRS sensitivity is moderate (60 %), because of its intrinsic detection limits, which could delay the diagnosis or lead to inappropriate therapy.

The use of somatostatin agonists (DOTATOC, DOTATATE, DOTANOC), radiolabeled with gallium-68 (68Ga) enables targeting of Somatostatin receptors (SSTRs) with a PET resolution. This has improved diagnosis of TNE with a gain in sensitivity of over 20% compared to SRS. Furthermore, patient irradiation and imaging protocol are significantly reduced.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18,

  * Patient with one of the following situations : suspicion of GEP, initial staging of non-metastatic GEP, GEP with unknown primary tumor, Restaging of GEP justifying focused therapeutic approach
  * Reference imaging within the last 3 months: multiphasic thoracoabdominal CT scan, liver MRI and SRS (SPECT/CT).

Exclusion Criteria:

* Pregnant or breast-feeding woman
* Other cancer disease
* GEP with grade 3 tumours
* Non GEP TNE (paragangliome, medullar thyroid cancer)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-04-22 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
interest of the realization of 68Ga-DOTATATE PET-CT in the detection of tumor sites in TNE diagnosis, staging and restaging | 12-15 months

SECONDARY OUTCOMES:
therapeutic impact of 68Ga-DOTATATE PET-CT in addition to reference imaging (SRS, CT, MRI): we will document the rate of changes in treatment options induced by PET-CT | 12-15 months

OTHER OUTCOMES:
therapeutic impact of 68Ga-DOTATATE PET-CT in addition to reference imaging (SRS, CT, MRI): we will document the rate of changes in treatment options induced by PET-CT | 12-15 months

CONTACTS AND LOCATIONS:
Overall Officials: David TAIEB, MD, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France